CLINICAL TRIAL: NCT04404335
Title: The Role of Anti-inflammatory Cytokines and Antimicrobial Peptide LL-37 Biomarkers in the Treatment of Periodontal Disease.
Status: Completed | Type: Observational
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, David Madruga-Gonzalez, Associate Professor, Universidad Rey Juan Carlos
Other Study IDs: LL-37PERIOURJC
Record Dates: First submitted 2020-05-17; First posted 2020-05-27 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: Antimicrobial peptides; Defensines; LL-37; Periodontal disease; Crevicular fluid; IL-4; IL-6; IL-10
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy (control group): This group will include a total of 30 patients free of periodontitis Samples of crevicular fluid to quantity levels of antimicrobial peptide LL-37 will be taken at baseline
  ELISA analysis of all samples will be performed by using a specific ELISA kit commercially available for human LL-37 and also IL-4, IL-6 and IL-10
  Interventions: Diagnostic Test: Crevicular fluid analysis by using ELISA testing.
- Periodontitis (test group): 30 Periodontal patients (subdivided in 2 groups of 15, depending of the severity of their disease):
  * 15 patients with Stage I-II periodontitis (mild/moderate)
  * 15 patients with Stage III-IV periodontitis (severe).
  Two sets of samples of crevicular fluid will be obtained before and after receiving a course of routine basic periodontal treatment (root scaling and planing).
  A reevaluation visit to re-assess clinical periodontal parameters will take place at 4-6 weeks after treatment. New samples of crevicular fluid will then be taken at this stage to compare the level of LL-37 before and after the treatment.
  ELISA analysis of all samples will be performed by using a specific ELISA kit commercially available for human LL-37 (HyCult Biotechnology, Uden, the Netherlands).
  Interventions: Diagnostic Test: Crevicular fluid analysis by using ELISA testing.

INTERVENTIONS:
Diagnostic Test: Crevicular fluid analysis by using ELISA testing. — Samples of crevicular fluid (fluid existing in the space between the gums and the roots of the teeth) will be obtained from healthy and periodontal patients. In periodontal patients, samples will be taken before and after receiving a routine course of periodontal treatment (root scale and polish) to assess the levels of a peptide called LL-37 and inflammatory cytokines (IL-4, IL-6, IL-10): Samples will then be analysed using laboratory procedures (ELISA)

SUMMARY:
Periodontal disease is an infectious pathology that consists of the destruction of the gums and supporting structures around the teeth. There are several mechanisms involved in this process. In healthy conditions there is a balance between the bacteria present in the gums and the defence mechanisms of the host to fight the disease. One of the substances involved in favouring this protective mechanism is a peptide called LL-37.

The aim of this study is to find out more about the rol of this peptide during this process by using a non invasive method of analysis consisting of analysing some samples of the fluid existing between the gums and the teeth.

This clinical study will take place at the University Clinic at the University Rey Juan Carlos, Alcorcon (Madrid), Spain. Patients that attend the clinic suffering from gum disease will be offered the possibility to participate in this study. A full questionnaire indicating the risks and benefits of participating in the study as well as the management of confidential personal data will be discussed with the participants in full detail. Full consent will be sought before commencing the study.

Firstly, all participants will receive a through periodontal (gum) examination to assess if they suffer from periodontal disease and to what extent (severity). Based on this preliminary data, patients will be classified in different categories.

Patients will be divided in two groups:

* 30 Healthy patients (no signs of periodontitis)
* 30 Periodontal patients (subdivided in 2 groups of 30, depending of the severity of their disease:

  * 15 patients with Stage I-II periodontitis (mild/moderate)
  * 15 patients with Stage III-IV periodontitis (severe).

The intervention will consist on taking samples of crevicular fluid (the fluid found in the space between the gum and the root of the tooth) to quantify the presence of LL-37 as well as IL-4, IL-6, IL-10, which seems to be associated with the defence mechanisms (immunity) of the host against periodontal disease. These samples will be analysed in the laboratory by using some specific procedure called ELISA.

All patients from the test group will receive a basic course of periodontal treatment (root scale and polish), which is intended to remove the bacteria causing the disease from the space between the gums and the roots (periodontal pocket). Samples of crevicular fluid will be obtained before commencing the treatment. After 4-6 weeks, a new periodontal examination will take place to assess if there is an improvement of the condition and also to quantify the levels of LL-37, IL-4, IL-6, IL-10.

The findings of this study will help to understand the role of this peptide in the defence mechanism of the host against periodontal disease. This could ultimately serve to develop new therapies that could include the use of this peptide in addition to the routine periodontal treatment prescribed to improve the healing conditions of the patient against periodontal disease.

DETAILED DESCRIPTION:
'The role of anti-inflammatory cytokines and antimicrobial peptide LL-37 biomarkers in the treatment of periodontal disease.

1. Introduction

   Periodontal disease is an infectious process that consists of the destruction of the supporting anatomical structures of the tooth, as a consequence of the inflammatory response to the periopathogenic activity of the subgingival bacterial plaque, which leads to an innate, inflammatory and adaptative immune response.

   The clinical manifestation of the disease depends of host and environmental factors as well as the specific microbiological agent involved. The interrelation amongst bacteria and the immunodefence mechanisms of the host constitute the base of the immunopathological mechanisms that lead to the disease. In healthy conditions, there is a balance between the activity of the periodontal microbiota and the host immune response.

   In the innate defence system of the oral cavity there are several antimicrobial peptides involved, being one of them, the human cathelicidin LL-37.

   The activity of antimicrobial peptides such as LL-37 in the gingival sulcus is considered one of the greatest defence mechanisms of the periodontum. The gingival epithelium not only constitutes a physical barrier to avoid bacterial invasion. Neutrophils migrate to the junctional epithelium and create a barrier between the bacterial plaque and the underlaying epithelium. They also produce antimicrobial peptides, one of them the 18 kDa (hCAP18). Once the neutrophils are activated in response to the bacterial aggression the release LL-37, with a similar activity to a broad-spectrum antibiotic.

   The total absence of this peptide (LL-37) has been associated to aggressive periodontitis, in particular in patients with a neutrophil deficiency such as those who suffer Morfan Kosmann syndrome

   The nature of this research aims to elucidate the role of LL-37 in periodontal disease by comparing the use of a none invasive technique such as crevicular fluid samples in patients that suffer periodontal disease, before and after receiving a course of basic periodontal treatment (root scaling and planing). In additionto the above, pro and antiinflammatory cytokines (IL-6, IL-4, IL-10 in particular) will also be evaluated before and after periodontal treatment. Samples obtained will be analysed by immunohystochemical analysis (ELISA). The quantification of LL-37 before and after periodontal treatment associated with the clinical findings observed may serve as diagnostic biomarker of the immunopathological response inherent to the periodontal disease.
2. Justification of research question. Current status

   Over the last years, a great effort by scientific community has been made in order to try to understand the complex immunopathological processes related to periodontal disease and the relationship between the activity of the periodontal microbiota and the host defence mechanisms.

   The relevance of this research may serve to understand in more detail the role of the antimicrobial peptide LL-37 in periodontal disease not only due to their bactericidal effect but in the modulation of the immunological response of the host and its activity before and after periodontal treatment. The lack of studies on this matter reflects the need for further research on this topic.

   Ultimately, the findings of this research may form the basis of a new therapeutic approach based on the use of LL-37 to help modulate the immunological response of the host in combination with conventional periodontal treatment. This may be particularly relevant in patients susceptible to develop periodontal or periimplant diseases or in particular cases that are resistant to conventional treatment alternatives.
3. Summary of intended research

The main aim of the study is to investigate the role of LL-37 in the immunopathological response of the periodontum. Subsequent aims are to investigate the possibility of using this microbial peptide to serve as diagnostic, prognostic as well as a therapeutic agent in the treatment of periodontal disease.

Research hypothesis: There are significant quantitative differences in the levels of LL-37 before and after periodontal treatment, with a significant reduction of LL-37 at re-evaluation (4-6 weeks after a course of basic periodontal treatment -root scaling and planing).

Null hypothesis: There are no significant quantitative differences in the levels of LL-37 before and after periodontal treatment

The objectives of the present study are:

1. Determine if healthy patients and patients with periodontal disease have different levels of LL-37, IL-6, IL-4 and IL-10 in crevicular fluid at baseline and related them to the stage/severity of periodontal disease.
2. Evaluate if after a course of basic periodontal treatment these levels of LL-37, IL-6, IL-4 and IL-10 at baseline are similar to the quantified levels on healthy patients at baseline.
3. With respect to crevicular fluid samples, evaluate if levels of LL-37, IL-6, IL-4 and IL-10 in teeth affected by periodontal disease differ from healthy sites on the same individual or if there are no significant differences in the above before and after a course of periodontal treatment.
4. Stablish a non-invasive protocol to evaluate the immunological state of the patient before and after periodontal treatment as prognostic factor.

4. Material and methods

Ethical approval from the Ethical Commite of University Rey Juan Carlos of Madrid (URJC) has been granted. A selection of patients of the "Master in Advanced Implantology, Tissue Regeneration and Implant supported prosthesis" of the FCU-URJC that fulfil the inclusion criteria and that consent to be part of the study will be made.

The criteria for entry were as follows: aged 18 or over, with no previous history of periodontal treatment in the last six months, and no medical or dental history that could contraindicate periodontal treatment. Exclusion criteria included current pregnancy or lactation, immunological disorders, periodontal treatment within the last 6 months, oral contraception and antibiotic usage within the last 3 months, infections (such as HIV, hepatitis, and tuberculosis). In addition, third molar teeth were excluded from GCF sampling for being often impacted or extracted

Smoker patients will not be excluded and will be classified as light smokers (less than 10 cigarettes/day) or heavy smokers (more than 10 cigarettes /day).

Diabetic patients will not be excluded either but will be identified and accounted for.

All patients included in the study will go through the following stages:

1. Complete periodontal examination (probing depth (PD), clinical attachment level (CAL), plaque index (PI), blood on probing (BOP)).
2. Patients will be divided in two groups:

   * 30 healthy patients (control)
   * 30 periodontal patients (test- periodontitis stage I-II (15 patients), periodontitis stage III- IV (15 patients).

Due to lack of in vivo studies, simple sample size calculation was made using a conservative power analysis (G*Power 3.1.9.4 program, 2009). The simple size (27 subjects) was based on a two-tailed test with an effective size of 0.05, an alphabetical error probability of 0.05, difference of 50% in mean value, standard deviations to be maxium 80% of the mean values and a power of 0.90.

Taking into account these parameters, a simple sample size between 21-30 patients per group is estimated.

Crevicular fluid samples will also be obtained following the manufacturers protocol using perio papers (Periopaper, Applied Biosystems, Inc, Foster City, CA). Teeth to be examined will be isolated with cotton rolls and air dried. Paper strips will be introduced into the gingival sulcus for approximately 30 seconds. Test group patients' samples will be taken from periodontally pathogenic sites and healthy sites. Heavily contaminated samples with saliva or blood will be discarded.

Samples will be stored at -80 C at the laboratory of Departamento de Ciencias Básicas de la Salud, Edificio Departamental I, Fundación Clínica Universitaria, URJC (Alcorcon). Once all samples are obtained, ELISA analysis of all samples will be performed by using a specific ELISA kit commercially available for human LL-37 (HyCult Biotechnology, Uden, the Netherlands) and commercially available kits for IL-4, IL-4, IL-6 and IL-10 ((Diaclone SAS; Besançon, France; 850.890, 950.035 and 850.880, respectively).

Patients of the test group will receive a course of basic periodontal treatment (root scaling and planing) and oral hygiene instructions after the first sample collection.

A re-evaluation appointment at 4-6 weeks will take place where new crevicular fluid samples of both groups will be obtained (test and control), to evaluate any statistically significant difference with respect to the quantity of LL-37 in relation to the baseline measurements recorded. After that, samples will be scrutinised again by performing ELISA assays following the protocol described above.

Once all results are obtained, statistical analysis of the samples will be carried out.

ELIGIBILITY:
The criteria for entry were as follows: aged 18 or over, with no previous history of periodontal treatment in the last six months, and no medical or dental history that could contraindicate periodontal treatment. Exclusion criteria included current pregnancy or lactation, immunological disorders, periodontal treatment within the last 6 months, oral contraception and antibiotic usage within the last 3 months, infections (such as HIV, hepatitis, and tuberculosis). In addition, third molar teeth were excluded from GCF sampling for being often impacted or extracted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This clinical study will take place at the University Clinic at the University Rey Juan Carlos, Alcorcon (Madrid), Spain. Patients that attend the clinic suffering from gum disease will be offered the possibility to participate in this study. A full questionnaire indicating the risks and benefits of participating in the study as well as the management of confidential personal data will be discussed with the participants in full detail. Full consent will be sought before commencing the study.
  Patients will be divided in two groups:
  * 30 Healthy patients (no signs of periodontitis)
  * 30 Periodontal patients (subdivided in 2 groups of 15, depending of the severity of their disease:
    * 15 patients with Stage I-II periodontitis (mild/moderate)
    * 15 patients with Stage III-IV periodontitis (severe).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
LL-37 in crevicular fluid in healthy/periodontal patients. | At baseline for healthy (control) and periodontal (test) groups and at 4-6 weeks after treatment for test group
  Crevicular fluid samples will also be obtained following the manufacturers protocol using perio papers (Periopaper, Applied Biosystems, Inc, Foster City, CA). Samples will be stored at -80 C at the laboratory of Departamento de Epidemiología y Salud Pública, Edificio Departamental I, Fundación Clínica Universitaria, URJC (Alcorcon). Once all samples are obtained, appropriate transport will be arranged to the Department of Natural Sciences, Biomedical Sciences, Hendon Campus, Middlesex University of London. There ELISA analysis of all samples will be performed by using a specific ELISA kit commercially available for human LL-37 (HyCult Biotechnology, Uden, the Netherlands).

SECONDARY OUTCOMES:
Periodontal parameters | At baseline for healthy (control) and periodontal (test) groups and at 4-6 weeks after treatment for test group
  Probing depth (PD)
Probing depth (PD) | At baseline for healthy (control) and periodontal (test) groups and at 4-6 weeks after treatment for test group
  Assessment of the depth of the gingival sulcus by inserting a calibrated periodontal probe
Clinical attachment level (CAL) | At baseline for healthy (control) and periodontal (test) groups and at 4-6 weeks after treatment for test group
  Assessment of the soft tissue from the cemento enamel junction (CEJ) to the gingival margin
Plaque index (PI) | At baseline for healthy (control) and periodontal (test) groups and at 4-6 weeks after treatment for test group
  By using plaque diclosing tablets to assess levels of plaque/oral hygiene
Blood on probing (BOP) | At baseline for healthy (control) and periodontal (test) groups and at 4-6 weeks after treatment for test group
  Record of the presence of blood at the time of inserting the periodontal probe into the gingival sulcus

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universitaria Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
At present there is no consideration to share this data

REFERENCES:
- [Background] Davidopoulou S, Diza E, Sakellari D, Menexes G, Kalfas S. Salivary concentration of free LL-37 in edentulism, chronic periodontitis and healthy periodontium. Arch Oral Biol. 2013 Aug;58(8):930-4. doi: 10.1016/j.archoralbio.2013.01.003. Epub 2013 Feb 8. PMID 23778112
- [Background] Turkoglu O, Emingil G, Kutukculer N, Atilla G. Gingival crevicular fluid levels of cathelicidin LL-37 and interleukin-18 in patients with chronic periodontitis. J Periodontol. 2009 Jun;80(6):969-76. doi: 10.1902/jop.2009.080532. PMID 19485828
- [Background] Putsep K, Carlsson G, Boman HG, Andersson M. Deficiency of antibacterial peptides in patients with morbus Kostmann: an observation study. Lancet. 2002 Oct 12;360(9340):1144-9. doi: 10.1016/S0140-6736(02)11201-3. PMID 12387964
- [Background] de Haar SF, Hiemstra PS, van Steenbergen MT, Everts V, Beertsen W. Role of polymorphonuclear leukocyte-derived serine proteinases in defense against Actinobacillus actinomycetemcomitans. Infect Immun. 2006 Sep;74(9):5284-91. doi: 10.1128/IAI.02016-05. PMID 16926422
- [Background] Barros SP, Williams R, Offenbacher S, Morelli T. Gingival crevicular fluid as a source of biomarkers for periodontitis. Periodontol 2000. 2016 Feb;70(1):53-64. doi: 10.1111/prd.12107. PMID 26662482
- [Background] Kinney JS, Morelli T, Oh M, Braun TM, Ramseier CA, Sugai JV, Giannobile WV. Crevicular fluid biomarkers and periodontal disease progression. J Clin Periodontol. 2014 Feb;41(2):113-120. doi: 10.1111/jcpe.12194. Epub 2013 Dec 12. PMID 24303954
- [Background] McCrudden MT, Orr DF, Yu Y, Coulter WA, Manning G, Irwin CR, Lundy FT. LL-37 in periodontal health and disease and its susceptibility to degradation by proteinases present in gingival crevicular fluid. J Clin Periodontol. 2013 Oct;40(10):933-41. doi: 10.1111/jcpe.12141. Epub 2013 Aug 18. PMID 23952216
- [Background] Greer A, Zenobia C, Darveau RP. Defensins and LL-37: a review of function in the gingival epithelium. Periodontol 2000. 2013 Oct;63(1):67-79. doi: 10.1111/prd.12028. PMID 23931055
- [Background] Mallapragada S, Wadhwa A, Agrawal P. Antimicrobial peptides: The miraculous biological molecules. J Indian Soc Periodontol. 2017 Nov-Dec;21(6):434-438. doi: 10.4103/jisp.jisp_325_16. PMID 29551860
- [Background] Khurshid Z, Naseem M, Yahya I Asiri F, Mali M, Sannam Khan R, Sahibzada HA, Zafar MS, Faraz Moin S, Khan E. Significance and Diagnostic Role of Antimicrobial Cathelicidins (LL-37) Peptides in Oral Health. Biomolecules. 2017 Dec 5;7(4):80. doi: 10.3390/biom7040080. PMID 29206168
- [Derived] Madruga D, Garcia MM, Martino L, Hassan H, Elayat G, Ghali L, Ceballos L. Positive correlational shift between crevicular antimicrobial peptide LL-37, pain and periodontal status following non-surgical periodontal therapy. A pilot study. BMC Oral Health. 2023 May 28;23(1):335. doi: 10.1186/s12903-023-03023-w. PMID 37246231